CLINICAL TRIAL: NCT03928483
Title: Evaluation of a Commercial Program on Weight Loss and Health Outcomes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00085970
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: This single-armed trial will have one condition: the modified WW Food program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified WW Food program (Experimental): Participants will be assigned to a SmartPoints budget and number and types of ZeroPoint foods.
  Interventions: Behavioral: Modified WW Food program

INTERVENTIONS:
Behavioral: Modified WW Food program — Participants will receive a structured, holistic, behavioral weight management program that encourages development of healthy habits to help individuals eat healthier, move more, and shift to a more helpful mindset.

SUMMARY:
To examine weight loss and acceptability of a modified WW program. This study is designed to detect differences in weight loss at the end of 24 weeks of intervention.

DETAILED DESCRIPTION:
This trial is an examination of a modified WW food program. The intention is to document the acceptability and efficacy of the dietary plan over 24 weeks. Subjects will participate in a program similar to WW Freestyle and have access to study-specific weekly workshops and a suite of study-specific digital tools for tracking eating, activity, and weight. Within a WW program, participants are provided instructions on calculating points for the foods and beverages they eat and drink. This study will examine the impact of the modified WW food program on weight and fitness levels of adults with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75 years
* Body Mass Index (BMI) of 25 to 43
* Self-reported desire to lose weight
* Willing to discontinue any current over-the-counter (OTC) supplements not recommended/prescribed by physician, with the exception of multivitamins or other vitamin supplement
* Willing to follow recommendations required by study protocol
* Willing to include demographic information (e.g., ethnicity, income and education)
* Use of a personal iPhone on a daily basis
* Basic app skills
* Reliable home Wi-Fi access
* Ability to commit to attending up to 27 study visits in approximately 26 weeks

Exclusion Criteria

* Participants that are currently, or within the last 6 months, trying to lose weight by following guidelines (e.g., self-initiated programs) or a structured weight-loss program (e.g., at a medical center, university, commercial programs)
* Participants who were a member of WW within the past 12 months.
* Participants who are involved in any other research studies at this time (also, cannot join other research studies while in this study, over the next 6 months).
* Pregnant, nursing, or planning on becoming pregnant over the next 9 months.
* Weight loss of ≥ 5 kg in the previous 6 months.
* History of clinically diagnosed eating disorder.
* Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., orthopedic limitations, heart problems)
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months.
* Taking any prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qysmia, Contrave, etc.) with the exception of subjects on a stable dose of SSRIs for 6 months
* Diuretic use, unless taken on a regular, daily basis for hypertension and on a stable dose for at least 30 days
* Chronic/inflammatory gastrointestinal disorders (irritable bowel syndrome is acceptable).
* History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months.
* Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg
* Diagnosis of type 1 or type 2 diabetes
* Previous surgical procedure for weight loss.
* Major surgery within the previous 6 months.
* Presence of implanted cardiac defibrillator or pacemaker.
* History of cancer within past 5 years or current treatment for cancer (completely resected basal or squamous cell carcinoma acceptable if treatment completed more than 6 months prior to enrollment).
* Hospitalization for psychiatric disorders during the past 12 months
* Self-reported alcohol use > 7/week standard drinks for females and > 14/week for males or meets DSM-5 criteria for mild or greater, Alcohol Use Disorder
* Planning to relocate in the next 9 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
body weight change (kg) | baseline to six months
  average body weight change (kg) from baseline to six months

SECONDARY OUTCOMES:
3-month change in weight (kg) | baseline to 3-months
  average 3-month change in weight (kg)
3-month change in weight, as a percentage of start weight | baseline to 3-months
  3-month change in weight, as a percentage of start weight
6-month changes in body weight as a percentage of start weight | baseline to 6-months
  6-month changes in body weight as a percentage of start weight
changes in Body Mass Index (BMI) | baseline, 3-months and 6-months
  changes in Body Mass Index (BMI)
waist circumference | baseline, 3-months and 6-months
  change in waist circumference as measured at natural waist with a non-stretch tape measure.
flexibility | baseline, 3-months and 6-months
  change in flexibility as measured via standard sit-and-reach protocol
aerobic stamina | baseline, 3-months and 6-months
  change in aerobic stamina as measured with the 6-minute walk test
blood pressure | baseline, 3-months and 6-months
  change in blood pressure as measured by a blood pressure monitor
food cravings | baseline, 3-months and 6-months
  change in reported food cravings as measured by the FCI-II
happiness | baseline, 3-months and 6-months
  change in reported happiness as measured using the Oxford Happiness Questionnaire
sleep quality and duration: Pittsburgh Sleep Quality Index | baseline, 3-months and 6-months
  change in sleep quality and duration as measured by the Pittsburgh Sleep Quality Index
weight related quality of life: Impact of Weight Related Quality of Life- Lite (IWQOL-Lite) | baseline, 3-months and 6-months
  change in reported weight related quality of life as measured by the Impact of Weight Related Quality of Life- Lite (IWQOL-Lite)
subjective sensations of hunger | baseline, 3-months and 6-months
  change in subjective sensations of hunger as measured by the Hunger Visual Analog Scale
personal food assessment | baseline and 6-months
  changes in reported personal food assessment as measured by the Block Food Frequency Questionnaire
program satisfaction: WW generated satisfaction questionnaire | 3-months and 6-months
  program satisfaction as measured by the WW generated satisfaction questionnaire
health related quality of life: SF-36 | baseline, 3-months and 6-months
  changes in reported health related quality of life as measured through the SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No